CLINICAL TRIAL: NCT04661488
Title: Safety and Reliability of Artificial Intelligence Driven Symptom Assessment in Children and Adolescentes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ETMK Dnro: 68 /1801/2020
Record Dates: First submitted 2020-11-26; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-11

CONDITIONS: Artificial Intelligence; Triage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and adolescence
  Interventions: Device: AI driven triage-system

INTERVENTIONS:
Device: AI driven triage-system — AI driven triage-system

SUMMARY:
Digital health technologies (DHT) are increasingly developed to support healthcare systems around the world. However, they are frequently lacking evidence-based medicine and medical validation. There is considerable need in the western countries to allocate healthcare resources accurately and give the population detailed and reliable health information enabling to take greater responsibility for their health. Intelligent patient flow management system (IPFM, product name Klinik Frontline) is developed to meet these needs. In practice, IPFM is used for decision support in the triaging and diagnostic processes as well as automatizing the management of inflow of the patients. The core of the IPFM is a clinical artificial intelligence (AI), which utilizes a comprehensive medical database of clinical correlations generated by medical doctors.

The study population of this research consists of patients from the Paediatric Emergency Clinic of Turku University Hospital (TUH). Data will be gathered during 6 months of piloting, after which the results will be analysed. Anticipated number of patients to the study is minimum of 500 patients, with objective to be 1 000. When attending to the hospital, patients or their guardians will report their demographics, background information and symptoms using structured IPFM online form. Results obtained from IPFM are blinded from the healthcare professional and IPFM does not affect professional's clinical decision making. The data obtained from IPFM online form and clinical data from the emergency department and TUH will be analysed after the data collection. The main aim of the research is to validate the use of IPFM by evaluating the association of IPFM output with 1) urgency and severity of the conditions; and 2) actual diagnoses diagnosed by medical doctors. The main hypotheses of the research are that 1) IPFM is safe and sensitive in evaluating the urgency of the conditions of arriving patients at the emergency department and that 2) IPFM has sufficient correlation of differential diagnosis with actual diagnosis made by medical doctor.

ELIGIBILITY:
Inclusion Criteria:

* all patients at the emergency department with acute symptoms

Exclusion Criteria:

* Emergency situation

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children and adolescence of all ages and comorbidities
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Emergency severity index (ESI) | 1.12.2020-31.12.2021
  AI-driven automated analysis of triage urgency (ESI index) will be compared with the index estimated by healthcare professionals

SECONDARY OUTCOMES:
Primary diagnosis | 1.12.2020-31.12.2021
  AI-driven automated analysis of diagnosis will be compared with the diagnosis estimated by healthcare professionals

IPD SHARING:
Plan to Share IPD: No